CLINICAL TRIAL: NCT04766294
Title: Is the Severity of COVID-19 in Obese and Diabetic Patients Linked to High Serum Levels of MMP-7, MMP-9, TGF-β and PDGF Macrophage Activation Markers?
Brief Title: Macrophage Activation Markers in COVID-19 Patients
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahed Fathallah Fahmy, lecturer of Medical Microbiology & Immunology department -Faculty of medicine- Sohag university, Sohag University
Other Study IDs: Soh-Med-21-02-20
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aiming to find the relation between the severity of COVID-19 in diabetic and obese patients and the high serum levels of matrix metalloproteinase-7 (MMP-7),matrix metalloproteinase-9 (MMP-9), TGF-β and PDGF Macrophage Activation Markers

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) commonly occurs in COVID-19 patients who are diabetic and obese, ARDS is characterized by inflammation and pulmonary fibrosis mediated by cytokines and biomarkers released from activated alveolar macrophages, also cytokine storm may occurs leading to multiple organ failure. These sequelae of COVID-19 disease in obese and diabetic patients are attributed to elevated plasma lipopolysaccharide which is the main activator of M1 and M2 macrophages. chronic activation of macrophages leads to production of profibrotic markers as transforming growth factor-β (TGF-β), platelet-derived growth factor (PDGF), matrix metalloproteinase-7 (MMP7) and matrix metalloproteinase-9 (MMP9) which promote fibrogenesis. In this research, we measure circulatory alveolar macrophage activation markers in COVID-19 obese patients with type 1 and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Overweight patients with body mass index higher than 25 and obese patients with body mass index higher than 30 were selected to be included
* Type one and type two diabetes mellitus patients were also included

Exclusion Criteria:

-

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients admitted to isolation hospital in Sohag "Sohag teaching hospital".
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Measurement of matrix metalloproteinase-7 "MMP-7" serum level (pg/ml) as a biomarker of macrophage activation | MMP-7 is measured after admission of patients to isolation hospital along 7 days interval for 21 days, 3 plasma samples are collected on the 7th day of admission, day 14 and day 21
  ELISA "Enzyme linked immunosorbent assay" technique.
Measurement of matrix metalloproteinase-9 "MMP-9" serum level (pg/L) as a biomarker of macrophage activation | MMP-9 is measured after admission of patients to isolation hospital along 7 days interval for 21 days, 3 plasma samples are collected on the 7th day of admission, day 14 and day 21
  ELISA "Enzyme linked immunosorbent assay" technique.
Measurement of transforming growth factor B "TGF-B" serum level ( pg/ml) as a biomarker of macrophage activation | TGF-B is measured after admission of patients to isolation hospital along 7 days interval for 21 days, 3 plasma samples are collected on the 7th day of admission, day 14 and day 21
  ELISA "Enzyme linked immunosorbent assay" technique.
Measurement of platelet derived growth factor "PDGF" serum level (ng/ml) as a biomarker of macrophage activation | PDGF is measured after admission of patients to isolation hospital along 7 days interval for 21 days, 3 plasma samples are collected on the 7th day of admission, day 14 and day 21
  ELISA "Enzyme linked immunosorbent assay" technique.

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Fathallah, lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of medicine - sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided